CLINICAL TRIAL: NCT04813809
Title: A Prospective, Open, Non-comparative, Single-centre Investigation to Study the Effect of BARRIER® EasyWarm® Active Self-warming Blanket on Skin- and Body Core Temperatures in Healthy Volunteers
Brief Title: A Clinical Investigation With BARRIER® EasyWarm®
Acronym: EasyWarm01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EasyWarm01
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
Keywords: Body temperature; Healthy volunteers; EasyWarm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BARRIER EasyWarm (Experimental): This is an open, non randomised, single arm study
  Interventions: Device: BARRIER EasyWarm

INTERVENTIONS:
Device: BARRIER EasyWarm — Application of BARRIER EasyWarm for 10 hours. The treatment with the investigational device will be according to the instruction stated on the investigational device.

SUMMARY:
This investigation is a prospective, open, non-comparative, single-center investigation with the aim to investigate the effect of BARRIER EasyWarm active self-warming blanket on skin- and body core temperatures. The investigation will enroll approximately 20 healthy volunteers in one investigation site and each subject will be evaluated for up to 10 hours in one visit.

DETAILED DESCRIPTION:
This investigation is a prospective, open, non-comparative, single-center investigation with the aim to investigate the effect of BARRIER EasyWarm active self-warming blanket on skin- and body core temperatures.

The investigation will enroll approximately 20 healthy volunteers in one investigation site. Each subject will be evaluated for up to 10 hours in one visit on site. Body core- and skin reference temperatures will be established before applying the blanket. After reference temperature assessments, the BARRIER EasyWarm is positioned on the subject with the neckline at the collarbone. Skin temperatures will be assessed with an IR camera and body core temperatures will be assessed with an ear thermometer at 30 min, 1 hour, 2, 3, 4, 5, 6, 7, 8, 9, and 10 hours post blanket application. Subject perception of heat from the blanket will be assessed at 30 minutes, 5 hours and 10 hours post blanket application by means of a five graded question.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Adult males and females ≥ 18 years old
3. Able to maintain a supine position up to 10 hours.

Exclusion Criteria:

1. Diseases/medical treatments that affect normal body temperature control:

   I. Persons who have/have had thyroid disease or who are treated with medications affecting the thyroid hormones

   II. Persons being treated with medication affecting normal body temperature control, based on investigator judgement.
2. Impaired circulation/vascular disease
3. Impaired sensitivity/neuropathy
4. Active skin disease
5. Female with temperature variations due to menopause
6. Pregnancy or lactation at time of study participation.
7. Person not suitable for the investigation according to the clinician's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Skin temperature | 10 hours
  Relative change in average skin temperature (ºC)

SECONDARY OUTCOMES:
Skin temperature 1 | 30 minutes, and 1, 2, 3, 4, 5, 6, 7, 8, 9 hours
  Relative change in average skin temperature at 30 minutes, and 1, 2, 3, 4, 5, 6, 7, 8 and 9 hours (ºC). Assessed with an IR camera.
Skin temperature 2 | 30 minutes, and 1, 2, 3, 4, 5, 6, 7, 8, 9 and10 hours
  Maximum skin temperature at 30 minutes, and 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 hours (ºC). Assessed with an IR camera.
Skin temperature 3 | 30 minutes, and 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 hours
  Average skin temperature at 30 minutes, and 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 hours (ºC). Assessed with an IR camera.
Body Core Temperature 1 | 30 minutes, and 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 hours
  Body core temperature (ºC) at 30 minutes, and 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 hours. Assessed with an ear thermometer.
Body Core temperature 2 | 30 minutes, and 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 hours
  Relative change in body core temperature (ºC) at 30 minutes, and 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 hours compared to baseline. Assessed with an ear thermometer.
Heat perception | 30 minutes, 5 hours and 10 hours
  Five-point question related to perception of heat from the BARRIER EasyWarm. Assessed at 30 minutes, 5 hours and 10 hours post application. Scale: Cold, cool, not cool or warm, warm, hot.

CONTACTS AND LOCATIONS:
Locations (1):
- /Sahlgrenska University Hospital/Clinical Trial Center/Gothia Forum, Gothenburg, Sweden